CLINICAL TRIAL: NCT02333565
Title: Combination of Everolimus and Octreotide LAR in Aggressive Recurrent Meningiomas.
Acronym: CEVOREM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-09; 2014-003694-42 (EudraCT Number); RCAPHM14_0080 (Other: APHM)
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Meningiomas; Resistant Meningiomas
MeSH Terms: conditions — Meningioma | interventions — Everolimus; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combinaison everolimus and octreotide (Experimental)
  Interventions: Drug: Everolimus; Drug: Octreotide

INTERVENTIONS:
Drug: Everolimus
Drug: Octreotide

SUMMARY:
To determine if combination of everolimus and octreotide exert an anti-tumoral activity in recurrent and/or aggressive meningiomas growth with limited adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients ≥ 18 years old with no maximum limited of age
* Histologically proven meningioma grade II and III; grade I meningioma may also be included, if progression is documented (see criteria 3), particularly in case of skull base location
* Progression is defined on 2 different MRI as an increase of meningioma's surface ≥ 5% by 3 months period (i.e. an increase of 5% over 3 months, 10% over 6 months, 15% over 9 months…) or as the apparition of a new unequivocal neurological symptom related to the meningioma. We considered as a new unequivocal neurological symptom a new occurring neurological symptom as, for instance, hemiparesia, oculomotor nerve palsy, visual loss, facial nerve palsy, facial neuralgia, directly related to meningioma and suggesting meningioma growth with increase of meningioma compression on neurological structures despite no increasing size on MRIs.
* Patients must have failed surgery, and not amenable to a new curative intended surgery
* Patients must have failed radiotherapy and/or radiosurgery
* Prior chemotherapy is allowed, if progression under the cytotoxic agent is clearly documented. An interval of 4 weeks after the last administration of the cytotoxic agent is warranted. Number of prior chemotherapies is not limited.
* Patients who have given their written consent
* Patients affiliated to a social insurance regime
* Adequate bone marrow function as shown by: Absolute Neutrophil Count ≥ 1.5 x 109/L,
* Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Adequate liver function as shown by; serum bilirubin ≤ 1.5 x Upper Limit of Normal; International Normalized Ratio < 1.3; alanine aminotransferase and aspartate aminotransferase ≤ 2.5 x Upper Limit of Normal - Adequate renal function: serum creatinine ≤ 1.5 x Upper Limit of Normal - Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L and fasting triglycerides ≤ 2.5 x Upper Limit of Normal. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after dyslipidemia treatment initiation.

Exclusion Criteria:

* Patients with symptomatic lithiasis
* Contra indication to octreotide and everolimus
* Women of child-bearing age who are using no effective means of contraception
* Pregnant or breast-feeding women or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes
* Patients receiving other investigational agents or who received an investigative drug or therapy within the last 30 days.
* Known intolerance or hypersensitivity to octreotide, everolimus or other rapamycin (sirolimus, temsirolimus)
* Uncontrolled diabetes mellitus defined by HbA1c>8.5%
* Patients who have any severe and/or uncontrolled medical condition:

unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to inclusion, serious uncontrolled cardiac arrhythmia, active or uncontrolled severe infection, cirrhosis, chronic active hepatitis or chronic persistent hepatitis, severely impaired lung function (spirometry and Diffusing Capacity of the lung for carbon monoxide 50% or less of normal and O2 saturation 88% or less at rest on room air), active, bleeding diathesis

* Patients receiving chronic treatment with immunosuppressive agent
* Patients with a known history of HIV seropositivity
* Patients who have a history of another primary malignancy ≤ 3 years, with the exceptions of non-melanoma skin cancer, and carcinoma in situ of uterine cervix.
* Females patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
The Progression Free Survival rate | 36 months
  Measured by the number of individuals without progression disease at 6 months, according to Response Assessment in Neuro-Oncology criteria's.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux Marseille, Marseille, France